CLINICAL TRIAL: NCT01062490
Title: Clinical Phase II Trial to Evaluate the Safety and Efficacy of Treosulfan Based Conditioning Prior to Allogeneic Haematopoietic Stem Cell Transplantation in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Treosulfan Based Conditioning Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Joachim Baumgart, PhD, medac Gesellschaft für klinische Spezialpraeparate mbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-FludT.8/MDS
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Myelodysplastic Syndrome
Keywords: Treosulfan; MDS; allogeneic stem cell transplantation; leukemia; Conditioning
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treosulfan (Experimental): Patients with myelodysplastic syndrome, (MDS) according to WHO classification (< 20 % myeloblasts in peripheral blood or bone marrow at initial diagnosis) indicated for allogeneic transplantation
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — 14 g/m2/d, day -6 to -4
  Other Names: Ovastat

SUMMARY:
This is a multicenter, multinational, non-randomized, non-controlled open-label phase II trial to evaluate the safety and efficacy of treosulfan in a combination regimen with fludarabine as conditioning therapy prior to allogeneic stem cell transplantation (SCT) in patients with MDS.

The aim is to demonstrate a clinical benefit compared to historical data with intravenous busulfan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with myelodysplastic syndrome, (MDS) according to WHO classification (< 20 % myeloblasts in peripheral blood or bone marrow at initial diagnosis) indicated for allogeneic transplantation
2. Availability of an HLA-identical sibling donor (MRD) or HLA-identical unrelated donor (MUD) HLA-identity defined by the following markers: HLA-A, -B, -DRB1, DQB1.
3. Target graft size (unmanipulated) bone marrow: 2 to 10 x 106 CD34+ cells/kg BW recipient or at least 2 x 108 nucleated cells /kg BW or peripheral blood: 4 to 10 x 106 CD34+ cells/kg BW recipient
4. Age > 18 and < 60 years
5. Karnofsky Index > 80 %
6. Adequate contraception in female patients of child-bearing potential
7. Written informed consent

Exclusion Criteria:

1. 'Secondary' or therapy-related MDS with known history of exposure to cytotoxic alkylating drugs and/or radiation therapy
2. Previous AML-induction therapy with more than two courses (e.g. in case of blast excess)
3. Previous allogeneic transplantation
4. Severe concomitant illnesses / medical conditions (e.g. impaired respiratory and/or cardiac function)
5. Known and manifested malignant involvement of the CNS
6. Active infectious disease
7. HIV- positivity or active hepatitis infection
8. Impaired liver function (Bilirubin > upper normal limit; Transaminases > 3.0 x upper normal limit)
9. Impaired renal function (Creatinine-clearance < 60 ml/min; Serum Creatinine > 1.5 x upper normal limit).
10. Pleural effusion or ascites > 1.0 L
11. Pregnancy or lactation
12. Known hypersensitivity to treosulfan and/or fludarabine
13. Participation in another experimental drug trial within 4 weeks before study
14. Non-co-operative behaviour or non-compliance
15. Psychiatric diseases or conditions that might impair the ability to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2004-11; Primary Completion 2008-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Evaluation of engraftment | 4 years
Safety: Evaluation of CTC grade 3 and 4 adverse events between Day -6 and Day +28: hyperbilirubinemia and mucositis/stomatitis, veno-occlusive disease, seizures | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Tapani Ruutu, MD, Principal Investigator — Biomedicum Helsinki 2 C, POB 705, Turkholmankatu 8 C, FIN-00029 HUS Helsinki, Finland
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Ruutu T, Volin L, Beelen DW, Trenschel R, Finke J, Schnitzler M, Holowiecki J, Giebel S, Markiewicz M, Uharek L, Blau IW, Kienast J, Stelljes M, Larsson K, Zander AR, Gramatzki M, Repp R, Einsele H, Stuhler G, Baumgart J, Mylius HA, Pichlmeier U, Freund M, Casper J. Reduced-toxicity conditioning with treosulfan and fludarabine in allogeneic hematopoietic stem cell transplantation for myelodysplastic syndromes: final results of an international prospective phase II trial. Haematologica. 2011 Sep;96(9):1344-50. doi: 10.3324/haematol.2011.043810. Epub 2011 Jun 9. PMID 21659356